CLINICAL TRIAL: NCT06520397
Title: Evaluation of the Efficacy and Safety of Dual-targeted Therapy With Upadacitinib and Ustekinumab Versus Intensified Ustekinumab Therapy in Crohn's Disease Patients With an Insufficient Response to Standard-dose Ustekinumab: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Dual-targeted Therapy With Upadacitinib and Ustekinumab Versus Intensified Ustekinumab Therapy in Crohn's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei Wang, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024ZSLYEC-070
Record Dates: First submitted 2024-07-14; First posted 2024-07-25 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease
Keywords: Ustekinumab; Upadacitinib; Dual-target therapy; Intensified therapy; Endoscopic remission
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab; upadacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual-target Therapy Group (Experimental): Participants in this group will receive the standard maintenance dosage of Ustekinumab administered subcutaneously, combined with the addition of Upadacitinib administered orally.
  Interventions: Drug: Ustekinumab and Upadacitinib
- Intensified Ustekinumab Monotherapy Group (Active Comparator): Participants in this group will receive an additional induction dose of Ustekinumab administered intravenously, followed by maintenance therapy with Ustekinumab.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab and Upadacitinib — Participants in this group will maintain the original Ustekinumab regimen, receiving 90 mg administered subcutaneously every 8 weeks. In addition, they will receive Upadacitinib administered orally at a dosage of 45 mg daily for 12 weeks. After the 12-week period, the dosage of Upadacitinib will be adjusted based on patient condition and clinical judgment, continuing until the evaluation at week 16. Clinical efficacy of the dual-target therapy will be evaluated at week 16.
  Arms: Dual-target Therapy Group
Drug: Ustekinumab — Participants will receive an additional induction dose of Ustekinumab administered intravenously at 6 mg/kg at baseline. This will be followed by subcutaneous maintenance therapy of 90 mg every 4 weeks. Clinical efficacy will be evaluated at week 16.
  Arms: Intensified Ustekinumab Monotherapy Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of dual-target therapy (Ustekinumab combined with Upadacitinib) versus intensified Ustekinumab monotherapy in patients with Crohn's disease who have an inadequate response to standard doses of Ustekinumab. The main questions it aims to answer are:

Is dual-target therapy more effective than intensified Ustekinumab monotherapy in achieving endoscopic remission in Crohn's disease patients?

Is dual-target therapy as safe as intensified Ustekinumab monotherapy in terms of adverse events?

Participants will:

Receive either dual-target therapy (Ustekinumab combined with Upadacitinib) or intensified Ustekinumab monotherapy.

Attend regular clinic visits for monitoring and assessments. Complete questionnaires about their symptoms and quality of life. Undergo routine blood tests and endoscopic evaluations to assess disease activity.

Researchers will compare the dual-target therapy group to the intensified Ustekinumab monotherapy group to see if dual-target therapy is more effective in achieving endoscopic remission and is as safe in terms of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 70 years at baseline (week 0).
* Active Crohn's Disease: Participants must have active Crohn's disease at baseline, defined as: CDAI > 150 and Endoscopic activity with SES-CD > 6, or SES-CD > 4 (for isolated ileal disease), excluding the contribution of the stricture component (Excluding the stricture component ensures recruitment of patients with a better chance of improvement, given the primary endpoint is endoscopic remission), and at least one of the following: CRP > 10 mg/L (upper limit of normal on local assay), Fecal calprotectin (FC) > 250 μg/g, active disease confirmed by imaging.
* Prior Ustekinumab Treatment: Participants must have had primary non-response or secondary loss of response to TNFi, and have undergone at least 16-24 weeks of standard-dose ustekinumab treatment, but still have active CD.
* Consent and Compliance: Participants must be capable and willing to provide written informed consent and comply with the requirements of the study protocol.
* General Health: The principal investigator (or designee) must determine that the participant is in good general health based on medical history, laboratory test results, physical examination, chest X-ray (CXR), and 12-lead electrocardiogram (ECG) obtained during the screening period.

Exclusion Criteria:

* Allergies: Participants with known allergies to UPA or UST excipients or components.
* Colonic Neoplasia: Participants with untreated or unresolved high-grade dysplasia or colon cancer.
* Active Infections: Participants with active infections at screening or baseline, including but not limited to pneumonia, pyelonephritis, or herpes zoster, or those with evidence of chronic infections that make them unsuitable for the study as per the investigator's assessment.
* Surgical Intervention: Participants who currently require or are expected to require surgical intervention for CD during the study period.
* Thrombosis: Participants with thrombosis identified through limb venous Doppler ultrasound or D-dimer screening.
* Lymphoproliferative Disorders: Participants with a history of lymphoproliferative disorders, including lymphoma, or those with signs and symptoms indicative of possible lymphoproliferative disease such as lymphadenopathy and/or splenomegaly.
* Immunodeficiency: Participants with any known congenital or acquired immunodeficiency, including common variable immunodeficiency, HIV infection, or organ transplantation.
* Pregnancy: Female participants with a positive pregnancy test at screening or baseline (week 0).
* Lactation or Pregnancy Plans: Female participants who are breastfeeding or planning to become pregnant during the study.
* Substance Abuse: Participants with a history of drug abuse (defined as the use of any illicit drug) or alcohol abuse within 1 year prior to screening.
* Investigator's Discretion: Participants deemed unsuitable for the study by the investigator for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the endoscopic remission rate at week 16. | Week 16
  Endoscopic remission is defined as an SES-CD score of less than 3, with no individual variable subscore exceeding 1.

SECONDARY OUTCOMES:
Clinical response rate at week 16 | Week 16.
  Comparison of the clinical response rate (CDAI score reduction by ≥100 points from baseline, or CDAI score <150) between the UPA+UST group and the UST-M group at week 16.
Endoscopic response rate at week 16 | Week 16
  Comparison of the endoscopic response rate (defined as a reduction in SES-CD score by >50% from baseline, or for ileal-limited disease with a baseline SES-CD score ≥4, a reduction of at least 50%) between the UPA+UST group and the UST-M group.
Deep remission rate at week 16 | Week 16
  Comparison of the deep remission rate (defined as clinical remission and no ulcers on endoscopy, SES-CD score <3, with no individual variable subscore exceeding 1) between the UPA+UST group and the UST-M group.
Biochemical remission rate at week 16 | Week 16
  omparison of the biochemical remission rate (defined as CRP levels within the normal reference range) between the UPA+UST group and the UST-M group
Normalization rate of fecal calprotectin levels at week 16 | Week 16
  Comparison of the normalization rate of fecal calprotectin levels (defined as fecal calprotectin <200 μg/g) between the UPA+UST group and the UST-M group.
Normalization rate of intestinal wall thickness on ultrasound at week 16 | Week 16
  Comparison of the normalization rate of intestinal wall thickness on ultrasound (defined as intestinal wall thickness <3 mm) between the UPA+UST group and the UST-M group.
Health-related quality of life assessment using the Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 16 and around Week 52
  Evaluation of health-related quality of life using the Inflammatory Bowel Disease Questionnaire (IBDQ). Assessment of the average change in total IBDQ score from baseline at week 16 and around week 52. The IBDQ score ranges from 32 to 224, with higher scores indicating better quality of life.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at week 16. | Week 16
  The short-term safety of the treatment regimen will be evaluated by assessing the number of participants with treatment-related adverse events. Adverse events will be categorized and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The evaluation will occur at week 16.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 at week 52 | Around Week 52
  The long-term safety of the treatment regimen will be evaluated by assessing the number of participants with treatment-related adverse events at week 52. Adverse events will be categorized and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Wang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raine T, Danese S. Breaking Through the Therapeutic Ceiling: What Will It Take? Gastroenterology. 2022 Apr;162(5):1507-1511. doi: 10.1053/j.gastro.2021.09.078. Epub 2022 Jan 4. PMID 34995533
- [Background] Schultheiss JPD, Mahmoud R, Louwers JM, van der Kaaij MT, van Hellemondt BP, van Boeckel PG, Mahmmod N, Jharap B, Fidder HH, Oldenburg B. Loss of response to anti-TNFalpha agents depends on treatment duration in patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2021 Nov;54(10):1298-1308. doi: 10.1111/apt.16605. Epub 2021 Sep 24. PMID 34559428
- [Background] Noor NM, Lee JC, Bond S, Dowling F, Brezina B, Patel KV, Ahmad T, Banim PJ, Berrill JW, Cooney R, De La Revilla Negro J, de Silva S, Din S, Durai D, Gordon JN, Irving PM, Johnson M, Kent AJ, Kok KB, Moran GW, Mowat C, Patel P, Probert CS, Raine T, Saich R, Seward A, Sharpstone D, Smith MA, Subramanian S, Upponi SS, Wiles A, Williams HRT, van den Brink GR, Vermeire S, Jairath V, D'Haens GR, McKinney EF, Lyons PA, Lindsay JO, Kennedy NA, Smith KGC, Parkes M; PROFILE Study Group. A biomarker-stratified comparison of top-down versus accelerated step-up treatment strategies for patients with newly diagnosed Crohn's disease (PROFILE): a multicentre, open-label randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 May;9(5):415-427. doi: 10.1016/S2468-1253(24)00034-7. Epub 2024 Feb 22. PMID 38402895
- [Background] Singh S, George J, Boland BS, Vande Casteele N, Sandborn WJ. Primary Non-Response to Tumor Necrosis Factor Antagonists is Associated with Inferior Response to Second-line Biologics in Patients with Inflammatory Bowel Diseases: A Systematic Review and Meta-analysis. J Crohns Colitis. 2018 May 25;12(6):635-643. doi: 10.1093/ecco-jcc/jjy004. PMID 29370397
- [Background] Parigi TL, D'Amico F, Abreu MT, Rubin DT, Dignass A, Dotan I, Jairath V, Magro F, Peyrin-Biroulet L, Ghosh S, Danese S. Difficult-to-treat inflammatory bowel disease: results from a global IOIBD survey. Lancet Gastroenterol Hepatol. 2022 May;7(5):390-391. doi: 10.1016/S2468-1253(22)00085-1. No abstract available. PMID 35397241
- [Background] Feagan BG, Sandborn WJ, Gasink C, Jacobstein D, Lang Y, Friedman JR, Blank MA, Johanns J, Gao LL, Miao Y, Adedokun OJ, Sands BE, Hanauer SB, Vermeire S, Targan S, Ghosh S, de Villiers WJ, Colombel JF, Tulassay Z, Seidler U, Salzberg BA, Desreumaux P, Lee SD, Loftus EV Jr, Dieleman LA, Katz S, Rutgeerts P; UNITI-IM-UNITI Study Group. Ustekinumab as Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2016 Nov 17;375(20):1946-1960. doi: 10.1056/NEJMoa1602773. PMID 27959607
- [Background] Adedokun OJ, Xu Z, Gasink C, Jacobstein D, Szapary P, Johanns J, Gao LL, Davis HM, Hanauer SB, Feagan BG, Ghosh S, Sandborn WJ. Pharmacokinetics and Exposure Response Relationships of Ustekinumab in Patients With Crohn's Disease. Gastroenterology. 2018 May;154(6):1660-1671. doi: 10.1053/j.gastro.2018.01.043. Epub 2018 Feb 1. PMID 29409871
- [Background] Ollech JE, Normatov I, Peleg N, Wang J, Patel SA, Rai V, Yi Y, Singer J, Dalal SR, Sakuraba A, Cohen RD, Rubin DT, Pekow J. Effectiveness of Ustekinumab Dose Escalation in Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2021 Jan;19(1):104-110. doi: 10.1016/j.cgh.2020.02.035. Epub 2020 Feb 26. PMID 32109634
- [Background] Haider SA, Yadav A, Perry C, Su L, Akanbi O, Kudaravalli P, Tripathi N, Hashim MA, Abdelsalam M, Hussein M, Elkheshen A, Patel V, Ali SE, Lamb L, Ingram K, Mayne C, Stuffelbeam AB, Flomenhoft D, Stromberg A, Barrett TA. Ustekinumab dose escalation improves clinical responses in refractory Crohn's disease. Therap Adv Gastroenterol. 2020 Oct 13;13:1756284820959245. doi: 10.1177/1756284820959245. eCollection 2020. PMID 33133239
- [Background] Bermejo F, Jimenez L, Algaba A, Vela M, Bastida G, Merino O, Lopez-Garcia A, Melcarne L, Rodriguez-Lago I, de la Maza S, Bouhmidi A, Barreiro-de Acosta M, Lopez-Serrano P, Carrillo-Palau M, Mesonero F, Orts B, Bonillo D, Granja A, Guerra I. Re-induction With Intravenous Ustekinumab in Patients With Crohn's Disease and a Loss of Response to This Therapy. Inflamm Bowel Dis. 2022 Jan 5;28(1):41-47. doi: 10.1093/ibd/izab015. PMID 33528018
- [Background] Privitera G, Pugliese D, Lopetuso LR, Scaldaferri F, Neri M, Guidi L, Gasbarrini A, Armuzzi A. Novel trends with biologics in inflammatory bowel disease: sequential and combined approaches. Therap Adv Gastroenterol. 2021 Apr 27;14:17562848211006669. doi: 10.1177/17562848211006669. eCollection 2021. PMID 33995579
- [Background] Yang E, Panaccione N, Whitmire N, Dulai PS, Vande Casteele N, Singh S, Boland BS, Collins A, Sandborn WJ, Panaccione R, Battat R. Efficacy and safety of simultaneous treatment with two biologic medications in refractory Crohn's disease. Aliment Pharmacol Ther. 2020 Jun;51(11):1031-1038. doi: 10.1111/apt.15719. Epub 2020 Apr 24. PMID 32329532
- [Background] Gold SL, Steinlauf AF. Efficacy and Safety of Dual Biologic Therapy in Patients With Inflammatory Bowel Disease: A Review of the Literature. Gastroenterol Hepatol (N Y). 2021 Sep;17(9):406-414. PMID 34602905
- [Background] Penagini F, Lonoce L, Abbattista L, Silvera V, Rendo G, Cococcioni L, Dilillo D, Calcaterra V, Zuccotti GV. Dual biological therapy and small molecules in pediatric inflammatory bowel disease. Pharmacol Res. 2023 Oct;196:106935. doi: 10.1016/j.phrs.2023.106935. Epub 2023 Sep 23. PMID 37748559
- [Background] Feng Z, Kang G, Wang J, Gao X, Wang X, Ye Y, Liu L, Zhao J, Liu X, Huang H, Cao X. Breaking through the therapeutic ceiling of inflammatory bowel disease: Dual-targeted therapies. Biomed Pharmacother. 2023 Feb;158:114174. doi: 10.1016/j.biopha.2022.114174. Epub 2022 Dec 31. PMID 36587559
- [Background] Fenster M, Alayo QA, Khatiwada A, Wang W, Dimopoulos C, Gutierrez A, Ciorba MA, Christophi GP, Hirten RP, Ha C, Beniwal-Patel P, Cohen BL, Syal G, Yarur A, Patel A, Colombel JF, Pekow J, Ungaro RC, Rubin DT, Deepak P. Real-World Effectiveness and Safety of Tofacitinib in Crohn's Disease and IBD-U: A Multicenter Study From the TROPIC Consortium. Clin Gastroenterol Hepatol. 2021 Oct;19(10):2207-2209.e3. doi: 10.1016/j.cgh.2020.10.025. Epub 2020 Oct 14. PMID 33068786
- [Background] Stalgis C, Deepak P, Mehandru S, Colombel JF. Rational Combination Therapy to Overcome the Plateau of Drug Efficacy in Inflammatory Bowel Disease. Gastroenterology. 2021 Aug;161(2):394-399. doi: 10.1053/j.gastro.2021.04.068. Epub 2021 May 4. No abstract available. PMID 33961886
- [Background] Loftus EV Jr, Panes J, Lacerda AP, Peyrin-Biroulet L, D'Haens G, Panaccione R, Reinisch W, Louis E, Chen M, Nakase H, Begun J, Boland BS, Phillips C, Mohamed MF, Liu J, Geng Z, Feng T, Dubcenco E, Colombel JF. Upadacitinib Induction and Maintenance Therapy for Crohn's Disease. N Engl J Med. 2023 May 25;388(21):1966-1980. doi: 10.1056/NEJMoa2212728. PMID 37224198
- [Background] Lee SD, Singla A, Harper J, Barahimi M, Jacobs J, Kamp KJ, Clark-Snustad KD. Safety and Efficacy of Tofacitinib in Combination With Biologic Therapy for Refractory Crohn's Disease. Inflamm Bowel Dis. 2022 Feb 1;28(2):309-313. doi: 10.1093/ibd/izab176. PMID 34347103
- [Background] Alayo QA, Khatiwada A, Patel A, Zulfiqar M, Gremida A, Gutierrez A, Rood RP, Ciorba MA, Christophi G, Deepak P. Effectiveness and Safety of Combining Tofacitinib With a Biologic in Patients With Refractory Inflammatory Bowel Diseases. Inflamm Bowel Dis. 2021 Oct 18;27(10):1698-1702. doi: 10.1093/ibd/izab112. No abstract available. PMID 34037225
- [Background] Alayo QA, Fenster M, Altayar O, Glassner KL, Llano E, Clark-Snustad K, Patel A, Kwapisz L, Yarur AJ, Cohen BL, Ciorba MA, Thomas D, Lee SD, Loftus EV Jr, Fudman DI, Abraham BP, Colombel JF, Deepak P. Systematic Review With Meta-analysis: Safety and Effectiveness of Combining Biologics and Small Molecules in Inflammatory Bowel Disease. Crohns Colitis 360. 2022 Feb 10;4(1):otac002. doi: 10.1093/crocol/otac002. eCollection 2022 Jan. PMID 35310082
- [Background] Yerushalmy-Feler A, Olbjorn C, Kolho KL, Aloi M, Musto F, Martin-de-Carpi J, Lozano-Ruf A, Yogev D, Matar M, Scarallo L, Bramuzzo M, de Ridder L, Kang B, Norden C, Wilson DC, Tzivinikos C, Turner D, Cohen S. Dual Biologic or Small Molecule Therapy in Refractory Pediatric Inflammatory Bowel Disease (DOUBLE-PIBD): A Multicenter Study from the Pediatric IBD Porto Group of ESPGHAN. Inflamm Bowel Dis. 2024 Feb 1;30(2):159-166. doi: 10.1093/ibd/izad064. PMID 37042978